CLINICAL TRIAL: NCT03824249
Title: Validation of Energy Expenditure Measurement With Indirect Calorimetry in Pediatric Patients Undergoing Non-invasive Ventilation Through a Single-limb Circuit With Intentional Leak: a Single Center, Cross-over, Non Pharmacological Study
Brief Title: Validation of Indirect Calorimetry in Children Undergoing Non-invasive Ventilation
Acronym: CALO-NIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/834
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2019-02

CONDITIONS: Respiratory Insufficiency in Children; Noninvasive Ventilation; Nutrition Assessment
Keywords: Energy Expenditure; Ventilator Weaning; Calorimetry, indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spontaneous breathing (Experimental): Performance of indirect calorimetry in spontaneously breathing children through the use of indirect calorimetry.
  Interventions: Diagnostic Test: Indirect Calorimetry
- NIV-CPAP (Experimental): Performance of indirect calorimetry in children undergoing Non-invasive continuous positive airway pressure (CPAP) of 4 centimeters of water (cmH2O). CPAP will be applied via single-limb circuit with intentional leak.
  Interventions: Diagnostic Test: Indirect Calorimetry
- NIV-PS (Experimental): Performance of indirect calorimetry in children undergoing Non-invasive continuous positive airway pressure (CPAP) of 4 cmH2O and Pressure support (PS) of 8 cmH2O. Non-invasive ventilation will be applied via single-limb circuit with intentional leak.
  Interventions: Diagnostic Test: Indirect Calorimetry

INTERVENTIONS:
Diagnostic Test: Indirect Calorimetry — Performance of indirect calorimetry in Canopy mode.
  Other Names: IC

SUMMARY:
Nutritional status in critically ill pediatric patients is considered a fundamental prognostic factor in terms of mortality, morbidity, complications and outcome. Many studies report how predictive equations most commonly applied are inaccurate, therefore under or over estimating the body energy requirements. For this reason, actual measurement of resting energy expenditure (REE) through indirect calorimetry (IC) is considered to be a better approach.

Currently, IC is not validated during the use of non-invasive ventilation.

Aim of the present study is to validate the measurement of REE with IC in pediatric patients undergoing non-invasive ventilation through a single-limb circuit with intentional leak.

ELIGIBILITY:
Inclusion Criteria:

* children admitted to the Pediatric Intensive Care Unit who completed the weaning phase from non-invasive ventilation.
* age ≤ 6 years
* patients whose parents provided signed informed consent

Exclusion Criteria:

* age > 6 years
* patients whose parents didn't provide signed informed consent

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure (REE) | 1 day
  Resting energy expenditure expressed in kcal/kg/die

SECONDARY OUTCOMES:
Carbon dioxide production (VCO2) | 1 day
  Quantity of carbon dioxide exhaled by the patients [expressed in ml/kg/min]
Oxygen consumption (VO2) | 1 day
  Quantity of oxygen consumed by the patients [expressed in ml/kg/min]
Respiratory quotient (RQ) | 1 day
  Respiratory quotient [expressed as VCO2/VO2]

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Langer, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano; Edoardo Calderini, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano; Carlo Agostoni, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy